CLINICAL TRIAL: NCT06356467
Title: Influence of Tumour and Patient's Related Factors on the Response to Medical Treatments in Well Differentiated GEP-NENs
Acronym: FARINET
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Gabriele Capurso, Professor, IRCCS San Raffaele
Other Study IDs: FARINET
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Neuroendocrine Tumors; GEP-NET
Keywords: GEP-NEN; NEN; GEP-NET
MeSH Terms: conditions — Neuroendocrine Tumors; Gastro-enteropancreatic neuroendocrine tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gastroenteropancreatic neuroendocrine neoplasms (GEP-NENs) represent the most common NeuroEndocrin Neoplasms (NEN) site, comprising 55-70% of all NENs, and they are extremely heterogeneous diseases in terms of clinical presentation and aggressiveness. In recent years there has been a significant increase in the incidence of such neoplasms, partially due to incidental findings of small indolent lesions. However, the behavior of GEP- NEN is variable and mainly dictated by some factors as age, sex, histologic grade, primary site, and stage at diagnosis1. As for grade which is defined by the proliferative activity as measured by mitotic count or ki67 staining, some 75% of neoplasms fall into the G1 grading category, 15% into the G2 category, and 10% into the G3 category. The probability of developing metastases is directly correlated with grading. In addition, the grading of GEP-NENs is also correlated with the type of differentiation of the neoplasm (well differentiated or poorly differentiated). Managing the complexity of this type of neoplasm has made it necessary to stratify patients into progression risk classes. The therapeutic approach is accordingly defined, and may include different treatments (surgery, loco-regional, targeted therapies, chemotherapies,...). Among treatments, the most widely used for patients with well-differentiated NENs are somatostatin analogs (SSAs), targeted therapies, and the combination of oral capecitabine and temozolomide. Systemic intravenous chemotherapy is instead employed in a subset of G3 neoplasms, especially if poorly differentiated.

DETAILED DESCRIPTION:
This is an observational retrospective multicentric cohort study. The primary outcome of the study is the global Progression-free survival (PFS) adjusted for the risk factors considered. In a subgroup of patients only previously enrolled in San Raffaele Hospital that were included in the BIO-PANCREAS study (approval number INT/96/2021, a local monocentric protocol in which blood and/or Endoscopic UltraSound-Fine Needle Aspiration (EUS-FNA) derived samples are collected for further molecular analyses), the trascriptome signature will also be investigated as potential biomarker of disease behavior. Retrospective enrolment will be performed from January 2015 to March 2023. As for the primary aim, patients' and tumours' related variables will be investigated as explanatory variables for the outcome "time to progression", hence this analysis will allow a response to the clinical question of whether these factors have an influence on tumour behavior under treatment. As for the subgroup analysis (analysis of trascriptome signatures), again, this will be investigated to test whether there is a signature able to discriminate different responses to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18
* Well-differentiated, localized (but not suitable for surgical treatment) or advanced (locally or with distant metastasis) GEP-NENs
* availability of data on site of primary tumor, stage of the, date of diagnosis
* treated with one (or more) of the following therapies:

  * Somatostatin analogs

    * G1 or G2 (Ki67 <10%) GEP-NENs
    * Treated for at least 6 months
    * first-line therapy (or as second-line after surgery in patients with residual disease or recurrence after surgical resection)
  * Sunitinib/Everolimus

    * G1/G2 GEP-NENs
    * Treated for at least 6 months
    * first- or second-line therapy
  * Capecitabine-Temozolomide (CAP-TEM)

    * G2 or G3 (Ki67 < 55%) GEP-NENs
    * first-, second-, or third-line therapy
    * Treated for at least 6 months

Exclusion Criteria:

* Age < 18aa
* Patients concomitantly treated with loco-regional treatments
* Patients previously treated with radioligand therapy
* Patients with need of CAP-TEM dose reduction of more than 33% for at least 3 administrations
* NENs of unknown primitivity (including patients with biopsy on secondary lesion compatible with metastasis from GEP-NEN, but with occult primary neoplasm)
* Patients with Mixed NENs (MiNENs)
* Patients with poorly differentiated neuroendocrine carcinoma
* Pregnancy and breastfeeding

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with well differentiated GEP-NENs
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Global Progression Free Survival (PFS) | 6 months
  Global pfs adjusted for the risk factors considered

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Capurso, PhD, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (1):
- IRCCS OSpedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No